CLINICAL TRIAL: NCT01563406
Title: Hub Cleansing to Prevent Hub Infection
Acronym: HUC-PHIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: U54CK000161-01W1 (NIH)
Record Dates: First submitted 2012-02-15; First posted 2012-03-27 (Estimated); Results first posted 2016-04-18 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2015-08

CONDITIONS: Bacteremia
Keywords: Needleless connectors; catheter hubs
MeSH Terms: conditions — Bacteremia | interventions — Ethanol; 2-Propanol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (4):
- Alcohol with 5 second scrub (Experimental): 70% isopropyl alcohol will be used to scrub catheter hubs for a duration of 5 seconds.
  Interventions: Other: 5 second scrub; Drug: 70% isopropyl alcohol
- Alcohol with 15 second scrub (Experimental): 70% isopropyl alcohol will be used to scrub catheter hubs for a duration of 15 seconds.
  Interventions: Other: 15 second scrub; Drug: 70% isopropyl alcohol
- Chlorhexidine with 5 second scrub (Experimental): 3.15% chlorhexidine/70% isopropyl alcohol will be used to scrub catheter hubs for a duration of 5 seconds.
  Interventions: Other: 5 second scrub; Drug: 3.15% chlorhexidine/70% isopropyl alcohol
- Chlorhexidine with 15 second scrub (Experimental): 3.15% chlorhexidine/70% isopropyl alcohol will be used to scrub catheter hubs for a duration of 15 seconds.
  Interventions: Other: 15 second scrub; Drug: 3.15% chlorhexidine/70% isopropyl alcohol

INTERVENTIONS:
Other: 15 second scrub — Scrub catheter hubs for 15 seconds before every access.
  Arms: Alcohol with 15 second scrub; Chlorhexidine with 15 second scrub
Other: 5 second scrub — Scrub catheter hubs for 15 seconds before every access.
  Arms: Alcohol with 5 second scrub; Chlorhexidine with 5 second scrub
Drug: 3.15% chlorhexidine/70% isopropyl alcohol — 3.15% chlorhexidine gluconate in 70% isopropyl alcohol pads will be used to disinfect catheter hubs prior to accessing central venous catheters during half of the study period.
  Other Names: Professional Disposables International Inc. Chlorascrub Swab
  Arms: Chlorhexidine with 15 second scrub; Chlorhexidine with 5 second scrub
Drug: 70% isopropyl alcohol — 70% isopropyl alcohol pads will be used to disinfect catheter hubs prior to accessing central venous catheters for the other half of the study period.
  Other Names: Professional Disposable International Inc Alcohol Prep Pad
  Arms: Alcohol with 15 second scrub; Alcohol with 5 second scrub

SUMMARY:
Central venous catheter infections are common preventable adverse events among hospital patients. Microbes may enter catheter hubs, also known as needleless connectors, and result in downstream contamination. This study aims to compare alcohol disinfection of catheter hubs to disinfection with chlorhexidine gluconate in alcohol, which has been proven to be a superior disinfectant at the site of central venous catheter insertion. Scrub duration of central venous catheter hubs will also be evaluated.

DETAILED DESCRIPTION:
A prospective randomized blinded crossover clinical trial will be performed in the medical intensive care unit at Rush University Medical Center. The intensive care unit will be divided into two regions (A&B). Hub disinfectants and duration of disinfection will be randomly assigned to these regions. After 1/2 of the study period, the agents will crossover, but the duration of scrubbing will remain the same, analogous to a 2 by 2 factorial design. Our primary endpoint will be internal contamination of hubs and catheters.

In February 2012 it was determined that the supplier of chlorhexidine and alcohol pads could not completely blind each pad. It was decided that a plain white sticker would be affixed to the front of each pad, but the safety information on the back of each pad would remain visible.

3/27/12-Internal hub contamination (yes/no)was clarified as the primary outcome.

On 5/10/12 a new sample size calculation adjusted the hub sample size needed to power the main effects based on more accurate information regarding the expected hub contamination rate. The expected hub contamination rate changed because of the more sensitive hub culture method that was adopted before the study began. This more sensitive method also allowed for a new secondary outcome of number of microbial colony forming units per hub.

The first crossover time selected was 6/11/12, prior to the midpoint of the study. This was done to try to improve a large imbalance in the group sizes.

On 6/11/12 a hold was placed on the catheter tip component of the study, because of an inability to collect tips.

On 8/7/12 the catheter tip outcome was dropped because of an inability to collect tips.

On 1/11/13 a second crossover was implemented in an effort to balance the sizes of the study groups.

ELIGIBILITY:
Inclusion Criteria:

* Medical intensive care unit patients with non-tunneled central venous catheters

Exclusion Criteria:

* Dialysis catheters
* Antibiotic-impregnated catheters
* Introducer sheaths
* Tunneled catheters

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2012-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary K Hayden, MD, Principal Investigator — Rush University Medical Center; Robert A Weinstein, MD, Principal Investigator — Cook County Health and Hospital Systems
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Rush University Medical Center adheres to the NIH Grant Policy on Sharing of Unique Research Resources including the Sharing of Biomedical Research Resources Principles and Guidelines for Recipients of NIH Grants and Contracts. Our response to requests for research resources from academic and other non-profit investigators will be timely and will be based on the Simple Letter Agreement for the Transfer of Materials as described in the Guidelines for Disseminating Research Resources Arising Out of NIH-Funded Research (Federal Register, Vol. 64, No 246, p.72094), and will not be more restrictive than the Uniform Biological Materials Transfer Agreement (UBMTA). Any intellectual property resulting from this study that can be patented will remain easily and widely available to the researchers in accordance with the NIH Principles and Guidelines. Distribution of resources to for-profit entities may occur under material transfer agreements or non-exclusive license arrangements.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 140 participants were recruited through 149 separate medical intensive care unit (MICU) admissions. Each MICU admission is treated as a separate enrollment.
Pre-assignment Details: Two separate wings of a 24-bed MICU were randomized to receive different intervention sequences. Wing A was assigned to a 15 sec scrub of 1) Alcohol; 2) chlorhexidine gluconate (CHG)+Alcohol; 3) Alcohol; and Wing B was assigned to a 5 sec scrub of 1) CHG+Alcohol; 2) Alcohol; 3) CHG+Alcohol.
Groups:
- Alcohol, 15 Second Scrub: - Description: Each catheter hub was disinfected before each access by scrubbing with 70% isopropyl alcohol alone for 15 sec
- Chlorhexidine+Alcohol, 15 Second Scrub: - Description: Each catheter hub was disinfected before each access by scrubbing with 3.15% chlorhexidine gluconate(CHG)/70% isopropyl alcohol for 15 sec
- Alcohol, 5 Second Scrub: - Description: Each catheter hub was disinfected before each access by scrubbing with 70% isopropyl alcohol alone for 5 sec.
- Chlorhexidine+Alcohol, 5 Second Scrub: - Description: Each catheter hub was disinfected before each access by scrubbing with 3.15% chlorhexidine gluconate(CHG)/70% isopropyl alcohol for 5 sec
Period: Overall Study
Arm/Group | Alcohol, 15 Second Scrub | Chlorhexidine+Alcohol, 15 Second Scrub | Alcohol, 5 Second Scrub | Chlorhexidine+Alcohol, 5 Second Scrub
Started | 60 (194 hubs) | 30 (102 hubs) | 30 (101 hubs) | 29 (112 hubs)
Completed | 60 (194 hubs) | 30 (102 hubs) | 30 (101 hubs) | 29 (112 hubs)
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 140 participants, 149 separate MICU admissions, 509 hubs total. Each MICU admission is treated as a separate enrollment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Alcohol, 15 Second Scrub | Chlorhexidine+Alcohol, 15 Second Scrub | Alcohol, 5 Second Scrub | Chlorhexidine+Alcohol, 5 Second Scrub | Total
Number analyzed (Participants) | 60 | 30 | 30 | 29 | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (17) | 61 (12) | 53 (17) | 59 (17) | 59 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 16 | 14 | 17 | 82
  Male | 25 | 14 | 16 | 12 | 67
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29 (9) | 31 (11) | 30 (14) | 32 (13) | 30 (11)
Mechanical ventilation [Number; unit: participants]
  Yes | 37 | 20 | 24 | 19 | 100
  No | 23 | 10 | 6 | 10 | 49
Decubitus ulcer [Number; unit: participants]
  Yes | 24 | 11 | 8 | 9 | 52
  No | 36 | 19 | 22 | 20 | 97
Diarrhea [Number; unit: participants]
  Yes | 20 | 16 | 13 | 12 | 61
  No | 40 | 14 | 17 | 17 | 88
Diabetes [Number; unit: participants]
  Yes | 21 | 13 | 8 | 7 | 49
  No | 39 | 17 | 22 | 22 | 100
Heart disease [Number; unit: participants]
  Yes | 32 | 16 | 12 | 21 | 81
  No | 28 | 14 | 18 | 8 | 68
Pulmonary Disease [Number; unit: participants]
  Yes | 14 | 6 | 8 | 8 | 36
  No | 46 | 24 | 22 | 21 | 113
Liver disease [Number; unit: participants]
  Yes | 5 | 4 | 2 | 3 | 14
  No | 55 | 26 | 28 | 26 | 135
Central venous catheter (CVC) type [Number; unit: hubs]
  Triple lumen | 135 | 69 | 61 | 86 | 351
  PICC | 59 | 33 | 40 | 26 | 158
Anatomic location of CVC [Number; unit: hubs]
  Internal/external jugular | 102 | 70 | 65 | 58 | 295
  Basilic/cephalic/brachial | 51 | 21 | 30 | 20 | 122
  Femoral | 21 | 11 | 6 | 21 | 59
  Subclavian | 18 | 0 | 0 | 13 | 31
  Unknown | 2 | 0 | 0 | 0 | 2
Time hub in place [Mean (Standard Deviation); unit: hours] | 95 (27) | 101 (41) | 100 (33) | 94 (25) | 97 (31)
No. hubs per patient [Median (Inter-Quartile Range); unit: hubs per patient] | 3 [2 to 3] | 3 [2 to 4] | 3 [2 to 3] | 3 [2 to 5] | 3 [2 to 4]

OUTCOME MEASURES:

1. Primary Outcome: Number of Central Venous Catheter Hubs With Internal Contamination
Description: This will be a qualitative outcome. It will be reported as "yes" or "no" for central venous catheter hub internal contamination. The number of hubs with internal contamination will be compared for the four study arms.
Time Frame: 15 months
Population: 140 participants were recruited through 149 separate medical intensive care unit (MICU) admissions. Each MICU admission is treated as a separate enrollment.
Measure: Number; unit: contaminated hubs
Units Other Than Participants: Hubs
Groups:
- Alcohol, 15 Second Scrub: Each catheter hub was disinfected before each access by scrubbing with 70% isopropyl alcohol alone for 15 sec.
- Chlorhexidine+Alcohol, 15 Second Scrub: Each catheter hub was disinfected before each access by scrubbing with 3.15% chlorhexidine gluconate(CHG)/70% isopropyl alcohol for 15 sec.
- Alcohol, 5 Second Scrub: Each catheter hub was disinfected before each access by scrubbing with 70% isopropyl alcohol alone for 5 sec.
- Chlorhexidine+Alcohol, 5 Second Scrub: Each catheter hub was disinfected before each access by scrubbing with 3.15% chlorhexidine gluconate(CHG)/70% isopropyl alcohol for 5 sec.
Arm/Group | Alcohol, 15 Second Scrub | Chlorhexidine+Alcohol, 15 Second Scrub | Alcohol, 5 Second Scrub | Chlorhexidine+Alcohol, 5 Second Scrub
Number analyzed (Participants) | 60 | 30 | 30 | 29
Number analyzed (Hubs) | 194 | 102 | 101 | 112
contaminated hubs | 42 | 18 | 39 | 14

2. Secondary Outcome: Number of Contaminated Central Venous Catheter Tips
Description: This will be a qualitative measure for central venous catheter tip contamination. The results will be reported as "yes" or "no".
Time Frame: 10 months
Population: Unable to collect a sufficient number of catheter tips to analyze. Therefore, this outcome was dropped early in the study.
Arm/Group | Alcohol, 15 Second Scrub | Chlorhexidine+Alcohol, 15 Second Scrub | Alcohol, 5 Second Scrub | Chlorhexidine+Alcohol, 5 Second Scrub
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Median Number of Microbial Colony Forming Units Per Hub Interior
Description: This will be a quantitative outcome. It will be reported as the median number of microbial colony forming units isolated per hub interior. The median number of microbial colony forming units isolated per hub interior will be compared for the four study arms.
Time Frame: 15 months
Measure: Median (Inter-Quartile Range); unit: colony forming units (CFU) per hub
Units Other Than Participants: Hubs
Arm/Group | Alcohol, 15 Second Scrub | Chlorhexidine+Alcohol, 15 Second Scrub | Alcohol, 5 Second Scrub | Chlorhexidine+Alcohol, 5 Second Scrub
Number analyzed (Participants) | 60 | 30 | 30 | 29
Number analyzed (Hubs) | 194 | 102 | 101 | 112
colony forming units (CFU) per hub | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 40] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: 15 months
Arm/Group | Alcohol, 15 Second Scrub | Chlorhexidine+Alcohol, 15 Second Scrub | Alcohol, 5 Second Scrub | Chlorhexidine+Alcohol, 5 Second Scrub
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/30 | 0/30 | 0/29
Other Adverse Events (participants affected / at risk) | 0/60 | 0/30 | 0/30 | 0/29

LIMITATIONS AND CAVEATS:
* Single MICU
* Large number of eligible hubs not evaluated
* Unbalanced hub collection among study arms
* Studied hub contamination only; unable to collect catheter tips
* Did not study central-line associated bloodstream infection itself

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No